CLINICAL TRIAL: NCT05089669
Title: Effects of an Interactive E-book to Enhance Nursing Students' Knowledge and Self-efficacy of Nursing Skill
Brief Title: Effects of an Interactive E-book to Enhance Nursing Skill
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: N202108014
Record Dates: First submitted 2021-09-26; First posted 2021-10-22 (Actual); Last update posted 2022-02-15 (Actual); Status verified 2021-09

CONDITIONS: Healthy
Keywords: Nursing students; Skill performance

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- interactive e-book (Experimental): The experimental group will read an interactive e-book for 90 minutes to learn nasogastric tube feeding.
  Interventions: Other: Interactive e-book
- comparison group (Active Comparator): The comparison group will read a paper textbook for 90 minutes to learn nasogastric tube feeding.
  Interventions: Other: paper textbook

INTERVENTIONS:
Other: Interactive e-book — The nasogastric tube feeding interactive e-book has a lot of elements such as text content, videos, pictures, links, and other interactive content with which the students can interact. The participants can use the interactive e-book to learn nasogastric tube feeding.
  Arms: interactive e-book
Other: paper textbook — The paper textbook has text content and pictures. The participants can use the paper textbook to learn nasogastric tube feeding.
  Arms: comparison group

SUMMARY:
It is necessary for nursing students to have sufficient knowledge and correct nursing skill before clinical practicum to provide patients appropriate care and improve nursing quality. The learning materials of nursing skills are mainly paper textbooks and handouts, which are one-way knowledge transmissions having limitations and deficiencies in nursing skill learning. Interactive e-books integrate multimedia such as text, images, and videos, which are more suitable for learning nursing skill and maximize the effectiveness of the learning materials. The present study aimed to develop a nasogastric tube feeding interactive e-book based on Information Processing Theory (IPT) and Attention, Relevance, Confidence, and Satisfaction Motivational Model (ARCS), hoping to improve students' learning motivation and learning effectiveness. This is a randomized controlled trial study. Convenience sampling will be applied. The participants will be recruited and randomly assigned into the experimental group and comparison group. The experimental group will read an interactive e-book to learn nasogastric tube feeding, while the comparison group will read a paper textbook.

DETAILED DESCRIPTION:
It is necessary for nursing students to have sufficient knowledge and correct nursing skill before clinical practicum to provide patients appropriate care and improve nursing quality. The learning materials of nursing skills are mainly paper textbooks and handouts, which are one-way knowledge transmissions having limitations and deficiencies in nursing skill learning. Interactive e-books integrate multimedia such as text, images, and videos, which are more suitable for learning nursing skill and maximize the effectiveness of the learning materials. In addition, the learning content can be updated at any time, in order that students can learn the latest skills and connect with clinical. The present study aimed to develop a nasogastric tube feeding interactive e-book based on Information Processing Theory (IPT) and Attention, Relevance, Confidence, and Satisfaction Motivational Model (ARCS), hoping to improve students' learning motivation and learning effectiveness. Therefore, the purpose of this study is to examine the effectiveness of using interactive e-book to enhance nursing students' knowledge and learning self-efficacy of nursing skill.

This is a randomized controlled trial study. Convenience sampling will be applied at a university in Northern Taiwan. It is expected that 60-100 participants will be recruited and randomly assigned into the experimental group and comparison group. The experimental group will read an interactive e-book to learn nasogastric tube feeding, while the comparison group will read a paper textbook. The questionnaires will be collected before the intervention, after the intervention, and after one month of the intervention. The questionnaires include demographic information, nasogastric tube feeding knowledge questionnaire, nasogastric tube feeding confidence scale, learning self-efficacy scale, nasogastric tube feeding skill test, and learning satisfaction questionnaire. This study will use SPSS 19.0 software for data analysis, including percentage, mean, standard deviation, t-test, chi-square test, and generalized estimation equation (GEE).

ELIGIBILITY:
Inclusion Criteria:

* students who major in nursing
* students have not yet learned nasogastric tube feeding skill.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2021-12-02 (Actual); Primary Completion 2022-01-21 (Actual); Study Completion 2022-01-21 (Actual)

PRIMARY OUTCOMES:
Nasogastric Tube Feeding Quiz | Baseline, before the intervention(T0)
  The Nasogastric Tube Feeding Quiz is a 15-item true/false questions with three responses (true, false, and not sure). Participants score 1 point for a correct answer and 0 for an incorrect answer or "not sure." The total score ranged 0-15 points. A higher score indicating a better knowledge of NG tube feeding.
Nasogastric Tube Feeding Quiz | Immediately following after the intervention(T1)
  The Nasogastric Tube Feeding Quiz is a 15-item true/false questions with three responses (true, false, and not sure). Participants score 1 point for a correct answer and 0 for an incorrect answer or "not sure." The total score ranged 0-15 points. A higher score indicating a better knowledge of NG tube feeding.
Nasogastric Tube Feeding Quiz | one month after the intervention(T2)
  The Nasogastric Tube Feeding Quiz is a 15-item true/false questions with three responses (true, false, and not sure). Participants score 1 point for a correct answer and 0 for an incorrect answer or "not sure." The total score ranged 0-15 points. A higher score indicating a better knowledge of NG tube feeding.
Confidence scale (C-scale) | Baseline, before the intervention(T0)
  A 5-item scale designed to measure participant's confidence level in performing a nursing skill. Each item had five responses and the total score ranged 5-25 points. A higher score indicating that nursing students felt more confident in performing the nursing skill.
Confidence scale (C-scale) | Immediately following after the intervention(T1)
  A 5-item scale designed to measure participant's confidence level in performing a nursing skill. Each item had five responses and the total score ranged 5-25 points. A higher score indicating that nursing students felt more confident in performing the nursing skill.
Confidence scale (C-scale) | one month after the intervention(T2)
  A 5-item scale designed to measure participant's confidence level in performing a nursing skill. Each item had five responses and the total score ranged 5-25 points. A higher score indicating that nursing students felt more confident in performing the nursing skill.
Learning Self-Efficacy Scale (L-SES) | Baseline, before the intervention(T0)
  A 12-item scale designed to measure student's learning self-efficacy for nasogastric tube feeding. Participants rate each item on a scale from 1 to 5. The total score ranged 12-60 points. A higher score indicating the nursing students have more confidence in their capability to learn nasogastric tube feeding.
Learning Self-Efficacy Scale (L-SES) | Immediately following after the intervention(T1)
  A 12-item scale designed to measure student's learning self-efficacy for nasogastric tube feeding. Participants rate each item on a scale from 1 to 5. The total score ranged 12-60 points. A higher score indicating the nursing students have more confidence in their capability to learn nasogastric tube feeding.
Learning Self-Efficacy Scale (L-SES) | one month after the intervention(T2)
  A 12-item scale designed to measure student's learning self-efficacy for nasogastric tube feeding. Participants rate each item on a scale from 1 to 5. The total score ranged 12-60 points. A higher score indicating the nursing students have more confidence in their capability to learn nasogastric tube feeding.
Nasogastric tube feeding skill test | three months after the intervention
  The Nasogastric tube feeding skill test is designed to test nasogastric tube feeding skill performance and competence. It requires participants to perform NG tube feeding in front of an examiner. The participants will be asked to demonstrate NG tube feeding in 10 minutes. The total score ranged 0-100 points. A higher score indicating the nursing students have a better ability of NG tube feeding.

SECONDARY OUTCOMES:
Satisfaction questionnaire | Immediately following after the intervention(T1)
  A 10-item scale designed to measure participant's level of satisfaction in learning materials. Participants rate each item on a scale from 1 (very dissatisfied) to 5 (very satisfied). The total score ranged 10-50. A higher score indicating high level of satisfaction in the learning materials.

CONTACTS AND LOCATIONS:
Overall Officials: Yeu-Hui Chuang, Principal Investigator — Taipei Medical University
Locations (1):
- Taipei Medical University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zuily S, Phialy L, Sevim E, Germain E, Unlu O, Dufrost V, Risse J, Clerc-Urmes I, Baumann C, Berman JR, Lockshin MD, Wahl D, Erkan D. Impact of antiphospholipid syndrome iBook on medical students' improvement of knowledge: An international randomized controlled study. Eur J Rheumatol. 2019 Sep 5;6(4):207-211. doi: 10.5152/eurjrheum.2019.19030. Print 2019 Oct. PMID 31657703
- [Background] Stirling A, Birt J. An enriched multimedia eBook application to facilitate learning of anatomy. Anat Sci Educ. 2014 Jan-Feb;7(1):19-27. doi: 10.1002/ase.1373. Epub 2013 May 6. PMID 23650104
- [Background] Payne KF, Goodson AM, Tahim A, Wharrad HJ, Fan K. Using the iBook in medical education and healthcare settings--the iBook as a reusable learning object; a report of the author's experience using iBooks Author software. J Vis Commun Med. 2012 Dec;35(4):162-9. doi: 10.3109/17453054.2012.747173. PMID 23278413
- [Background] Liu Y, Chou PL, Lee BO. Effect of an interactive e-book on nursing students' electrocardiogram-related learning achievement: A quasi-experimental design. Nurse Educ Today. 2020 Jul;90:104427. doi: 10.1016/j.nedt.2020.104427. Epub 2020 Apr 10. No abstract available. PMID 32311667
- [Background] Hsiao CC, Tiao MM, Chen CC. Using interactive multimedia e-Books for learning blood cell morphology in pediatric hematology. BMC Med Educ. 2016 Nov 14;16(1):290. doi: 10.1186/s12909-016-0816-9. PMID 27842530